CLINICAL TRIAL: NCT06691126
Title: Pharmacokinetic Study of Terpinolene in Healthy Subjects (PKT Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: Institute for Human Development and Potential (IHDP), Singapore (Other)
Responsible Party: Principal Investigator, Chun Yip James Chan, Principal Scientist I, Singapore Institute of Food and Biotechnology Innovation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-099
Record Dates: First submitted 2024-11-08; First posted 2024-11-15 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Pharmacokinetics of Terpinolene
MeSH Terms: interventions — terpinolene; Olive Oil

STUDY DESIGN:
Intervention Model Description: The study will be carried out as a single arm, unblinded, PK study. The total duration of the study is about 24 hours, excluding screening and enrolment time (up to 1 hour).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): n=15, single oral dose of 200mg of food-grade terpinolene in 5ml of olive oil
  Interventions: Other: Terpinolene in olive oil

INTERVENTIONS:
Other: Terpinolene in olive oil — Single oral dose of 200mg food-grade terpinolene in 5ml of olive oil

SUMMARY:
The study aims to check if our prediction about the uptake, distribution, and elimination of terpinolene (a food additive commonly found in e.g. fruits and herbs) from the human body is accurate.

DETAILED DESCRIPTION:
Traditionally, the toxicological hazards of chemical substances have been identified and evaluated using animal studies. With the global shift towards limiting the use of animals in human safety assessment, "Next Generation Risk Assessment (NGRA)" has been conceptualized as a human-relevant, exposure-led approach integrating in silico, in chemico and in vitro methodologies. Consequently, in silico physiologically based pharmacokinetic (PBPK) modelling strategies have emerged as a central component of the NGRA paradigm. By mapping compound behaviour (i.e. absorption, distribution, metabolism and excretion) in the body to a physiologically realistic compartmental structure comprising various organs connected by the circulating blood system, PBPK models (i) provide the link between in vitro hazard data and human-relevant exposures and (ii) enable conversion of external doses to internal exposures which can then be compared to internal thresholds of toxicological concern (iTTC).

Established methods exist to develop a PBPK model for any chemical based solely on in vitro and in silico parameters. However, assessment of the predictive accuracies of any PBPK model-derived simulations is highly reliant on the availability of in vivo pharmacokinetic (PK) datasets. This inherently limits the widespread applicability of PBPK modelling to the vast chemical space of non-pharmacological entities whereby there is a paucity of in vivo data. To circumvent this limitation, Ellison et al. introduced a read across framework for evaluating the PBPK model of a target chemical (chemical with no PK data) using PK data from an analogous source chemical (chemical with existing PK data).

In this study, the investigator aims to further evaluate and develop this PK read-across approach to consider non-pharmaceutical compounds. A target compound with no human PK data available was identified, which is a food flavouring agent, terpinolene and its source compound, limonene. A PBPK model for terpinolene will be built and used to compare the in vitro absorption, distribution, metabolism and elimination (ADME) parameters between terpinolene and limonene. To further validate this read-across approach, a prospective clinical study to obtain the missing in vivo PK of terpinolene is proposed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-50
* Chinese, Malay and Indian ethnicities
* Male or female
* Adequate fluency in the English language to understand the informed consent process, study instructions and study assessments
* Sufficient vision and hearing to complete the study procedures
* Willing and able to participate and to give written informed consent

Exclusion Criteria:

* Past (<3 months prior to the study) or current major metabolic, endocrine, gastrointestinal or cardiovascular disease
* Individuals diagnosed with non-alcoholic fatty liver disease
* Major surgery in the past 2 months
* On chronic medication
* Allergy to olive oil
* Vegetarian/vegan
* Smoking
* Pregnant or lactating
* Alcohol intake >1 units per day
* Body Mass Index <18.5 kg/m2 or ≥27 kg/m2
* Body weight <54 kg
* Member of the study team or their immediate family members

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Plasma terpinolene concentration | 24 hours
  Blood samples will be collected at 9 timepoints

CONTACTS AND LOCATIONS:
Overall Officials: James Chan, PhD, Principal Investigator — Singapore Institute of Food and Biotechnology Innovation (SIFBI), A*STAR
Locations (1):
- Human Development Research Centre, IHDP, A*STAR, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No